CLINICAL TRIAL: NCT00003492
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Large Cell, Undifferentiated Or Poorly Differentiated Stage IV Carcinoma of the Lung
Brief Title: Antineoplaston Therapy in Treating Patients With Stage IV Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066531; BC-LA-4 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Stage IV Lung Cancer
Keywords: Stage IV large cell lung cancer; Stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Stage IV Lung Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Stage IV Lung Cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage IV Pancreatic Cancer.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage IV Lung Cancer.

DETAILED DESCRIPTION:
Stage IV Lung Cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV Lung Cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV Lung Cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter. Cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed large cell, undifferentiated, or poorly differentiated stage IV lung cancer unlikely to have a curative response to existing standard regimens
* Measurable disease by MRI or CT scan

  * At least 2 cm in diameter

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal insufficiency
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections
* No other concurrent serious disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agent

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agent

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Recovered from prior surgery

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agent allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1996-04-10 (Actual); Primary Completion 2000-12-01 (Actual); Study Completion 2000-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with Stage IV Lung Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 9
Completed | 3
Not Completed | 6
Not completed — Not evaluable | 6

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 61.4 [45.8 to 74.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response or Stable Disease
Description: An objective response is a complete or partial response. A complete response is complete disappearance of all tumors by physical examination and radiographic studies for a minimum duration of four weeks. A partial response is > 50% reduction in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of four weeks. Stable disease indicates > 50% change in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of twelve weeks.
Time Frame: 16 months
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 3
Participants
  Stable Disease | 1
  Progressive Disease | 2

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Description: Nine patients were recruited between April 1996 and November 2000. All study subjects were seen at the Burzynski Clinic in Houston TX.
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 1
Lung (pneumonia) (Infections and infestations) | 1
Neuropathy: motor (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Rigors/chills (General disorders) | 1
Edema/Fluid retention (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Lung (pneumonia) (Infections and infestations) | 1
Other (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Hyperglycemia (Investigations) | 2
Hypernatremia (Investigations) | 6
Hypokalemia (Investigations) | 7
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 2
Pain: Head/headache (General disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No